CLINICAL TRIAL: NCT00760149
Title: Pharmacokinetics and Pharmacodynamics of High Versus Standard Dose Rifampicin in Patients With Pulmonary Tuberculosis in the Kilimanjaro Region, Tanzania.
Brief Title: Pharmacokinetics and Pharmacodynamics of High Versus Standard Dose Rifampicin in Patients With Pulmonary Tuberculosis
Acronym: High RIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Sanofi (Industry); Kilimanjaro Christian Medical Centre, Tanzania (Other); Kibong'oto National Tuberculosis Hospital, Sanya Juu, Tanzania (Unknown); University Centre for Chronic Diseases Dekkerswald, Groesbeek, The Netherlands (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Rob Aarnoutse, PharmD, PhD, Radboud University Nijmegen Medical Centre, the Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APRIORI 4.1; PACTR2009060001493909 (Registry Identifier: www.pactr.org)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; rifampicin; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): 50 patients, treated with the standard anti-TB regimen, including rifampicin (600 mg), isoniazid (300 mg), pyrazinamide (30 mg/kg), ethambutol (15 mg/kg), administered daily, orally, during the intensive phase of TB treatment. In addition they will receive 2 placebo tablets resembling rifampicin 300 mg.
  Interventions: Drug: Rifampicin in higher doses
- 2 (Active Comparator): 50 patients, treated with rifampicin (900 mg), and the other drugs in standard dosages (isoniazid (300 mg), pyrazinamide (30 mg/kg), ethambutol (15 mg/kg)), administered daily, orally, during the intensive phase of TB treatment. In addition they will receive 1 placebo tablet resembling rifampicin 300 mg.
  Interventions: Drug: Rifampicin in higher doses
- 3 (Active Comparator): 50 patients, treated with rifampicin (1200 mg), and the other drugs in standard dosages (isoniazid (300 mg), pyrazinamide (30 mg/kg), ethambutol (15 mg/kg)), administered daily, orally, during the intensive phase of TB treatment.
  Interventions: Drug: Rifampicin in higher doses

INTERVENTIONS:
Drug: Rifampicin in higher doses — Rifampicin 900 mg (study arm 2), and rifampicin 1200 mg (study arm 3)

SUMMARY:
In this phase II clinical trial, the pharmacokinetics, safety and (short-term) efficacy of higher than standard doses rifampicin will be studied during the intensive phase of tuberculosis (TB) treatment. Patients enrolled in this study will either get the standard TB regimen (including 600 mg rifampicin; first study arm), or 900 mg rifampicin plus isoniazid, ethambutol and pyrazinamide in standard dosages (second study arm), or 1200 mg rifampicin plus the other drugs in standard dosages (third study arm). All patients will get the standard TB regimen during the continuation phase of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a newly diagnosed pulmonary tuberculosis, confirmed by a positive smear of at least two sputum specimens with ZN staining.
* Participant is willing to be tested for HIV.
* Participant is at least 18, but not more than 65 years of age at the day of the first dosing of study medication.
* Participant is admitted to KNTH or KCMC during the intensive phase of TB treatment.
* Participant is able and willing to attend to KNTH or KCMC regularly during the continuation phase of TB treatment.
* Participant is able to understand and willing to sign the Informed Consent Form prior to screening evaluations.
* Female participants should understand that it is important not to get pregnant during the study. They should agree on taking measures to prevent them from getting pregnant during the study. They should agree on taking measures to prevent them from getting pregnant, such as using a contraceptive device or barrier method.

Exclusion Criteria:

* Participant has been treated with anti-tuberculosis drugs during the past three years.
* Participant's body weight is less than 50 kg.
* Participant has abnormal liver function test or serum creatinine (defined as levels higher than the upper limit of normal).
* Participant has a relevant medical history or current condition that might interfere with drug absorption, distribution, metabolism or excretion (i.e. chronic gastro-intestinal disease, Diabetes Mellitus, renal or hepatic disease, use of concomitant drugs that interfere with the pharmacokinetics of anti-TB drugs).
* Participant is on anti-retroviral treatment at inclusion.
* Participant has a CD4 count less than 350 cells/mm3.
* Participant has a Karnofsky score of less than 40.
* Participant is pregnant or breastfeeding.
* Participant has a Multi Drug Resistant (MDR)-TB for which another than the standard treatment regimen is needed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of rifampicin, desacetylrifampicin, isoniazid, pyrazinamide, ethambutol | Steady state, week 6

SECONDARY OUTCOMES:
Occurrence of adverse events | baseline, week 1, 2, 4, 6, 8, 10, 12
Bacteriological response of Mycobacterium tuberculosis | Almost daily during first 8 weeks
Compare accuracy of surrogate markers (SSCC, mRNA, cytokines) with standard two-month sputum conversion marker | Almost daily during first 8 weeks
Documenting the occurrence of mixed Mycobacterium tuberculosis strain infections | Almost daily during first 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob Aarnoutse, Pharm-D, PhD, Principal Investigator — Radboud University Medical Center; Gibson Kibiki, MD, MMed, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre,Moshi,Tanzania; Martin Boeree, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Center/UCCZ Dekkerswald
Locations (1):
- Kibong'oto National Tuberculosis Hospital, Sanya Juu, Kilimanjaro, Tanzania

REFERENCES:
- [Background] Frieden TR, Sterling TR, Munsiff SS, Watt CJ, Dye C. Tuberculosis. Lancet. 2003 Sep 13;362(9387):887-99. doi: 10.1016/S0140-6736(03)14333-4. PMID 13678977
- [Background] Iseman MD. Tuberculosis therapy: past, present and future. Eur Respir J Suppl. 2002 Jul;36:87s-94s. doi: 10.1183/09031936.02.00309102. PMID 12168751
- [Background] Ginsberg AM, Spigelman M. Challenges in tuberculosis drug research and development. Nat Med. 2007 Mar;13(3):290-4. doi: 10.1038/nm0307-290. No abstract available. PMID 17342142
- [Background] Mitchison DA. Role of individual drugs in the chemotherapy of tuberculosis. Int J Tuberc Lung Dis. 2000 Sep;4(9):796-806. PMID 10985648
- [Background] Diacon AH, Patientia RF, Venter A, van Helden PD, Smith PJ, McIlleron H, Maritz JS, Donald PR. Early bactericidal activity of high-dose rifampin in patients with pulmonary tuberculosis evidenced by positive sputum smears. Antimicrob Agents Chemother. 2007 Aug;51(8):2994-6. doi: 10.1128/AAC.01474-06. Epub 2007 May 21. PMID 17517849
- [Background] Jayaram R, Gaonkar S, Kaur P, Suresh BL, Mahesh BN, Jayashree R, Nandi V, Bharat S, Shandil RK, Kantharaj E, Balasubramanian V. Pharmacokinetics-pharmacodynamics of rifampin in an aerosol infection model of tuberculosis. Antimicrob Agents Chemother. 2003 Jul;47(7):2118-24. doi: 10.1128/AAC.47.7.2118-2124.2003. PMID 12821456
- [Background] Kreis B, Pretet S, Birenbaum J, Guibout P, Hazeman JJ, Orin E, Perdrizet S, Weil J. Two three-month treatment regimens for pulmonary tuberculosis. Bull Int Union Tuberc. 1976;51(1):71-5. No abstract available. PMID 1030315
- [Background] Long MW, Snider DE Jr, Farer LS. U.S. Public Health Service Cooperative trial of three rifampin-isoniazid regimens in treatment of pulmonary tuberculosis. Am Rev Respir Dis. 1979 Jun;119(6):879-94. doi: 10.1164/arrd.1979.119.6.879. PMID 110184
- [Background] Burman WJ, Gallicano K, Peloquin C. Comparative pharmacokinetics and pharmacodynamics of the rifamycin antibacterials. Clin Pharmacokinet. 2001;40(5):327-41. doi: 10.2165/00003088-200140050-00002. PMID 11432536
- [Background] Ruslami R, Nijland HM, Alisjahbana B, Parwati I, van Crevel R, Aarnoutse RE. Pharmacokinetics and tolerability of a higher rifampin dose versus the standard dose in pulmonary tuberculosis patients. Antimicrob Agents Chemother. 2007 Jul;51(7):2546-51. doi: 10.1128/AAC.01550-06. Epub 2007 Apr 23. PMID 17452486
- [Background] Ruslami R, Nijland H, Aarnoutse R, Alisjahbana B, Soeroto AY, Ewalds S, van Crevel R. Evaluation of high- versus standard-dose rifampin in Indonesian patients with pulmonary tuberculosis. Antimicrob Agents Chemother. 2006 Feb;50(2):822-3. doi: 10.1128/AAC.50.2.822-823.2006. No abstract available. PMID 16436757
- [Background] Solera J, Rodriguez-Zapata M, Geijo P, Largo J, Paulino J, Saez L, Martinez-Alfaro E, Sanchez L, Sepulveda MA, Ruiz-Ribo MD. Doxycycline-rifampin versus doxycycline-streptomycin in treatment of human brucellosis due to Brucella melitensis. The GECMEI Group. Grupo de Estudio de Castilla-la Mancha de Enfermedades Infecciosas. Antimicrob Agents Chemother. 1995 Sep;39(9):2061-7. doi: 10.1128/AAC.39.9.2061. PMID 8540716
- [Background] Kochar DK, Aseri S, Sharma BV, Bumb RA, Mehta RD, Purohit SK. The role of rifampicin in the management of cutaneous leishmaniasis. QJM. 2000 Nov;93(11):733-7. doi: 10.1093/qjmed/93.11.733. PMID 11077029
- [Background] Rosenthal IM, Williams K, Tyagi S, Peloquin CA, Vernon AA, Bishai WR, Grosset JH, Nuermberger EL. Potent twice-weekly rifapentine-containing regimens in murine tuberculosis. Am J Respir Crit Care Med. 2006 Jul 1;174(1):94-101. doi: 10.1164/rccm.200602-280OC. Epub 2006 Mar 30. PMID 16574936
- [Background] Fox W, Ellard GA, Mitchison DA. Studies on the treatment of tuberculosis undertaken by the British Medical Research Council tuberculosis units, 1946-1986, with relevant subsequent publications. Int J Tuberc Lung Dis. 1999 Oct;3(10 Suppl 2):S231-79. No abstract available. PMID 10529902
- [Background] Peloquin CA, Namdar R, Singleton MD, Nix DE. Pharmacokinetics of rifampin under fasting conditions, with food, and with antacids. Chest. 1999 Jan;115(1):12-8. doi: 10.1378/chest.115.1.12. PMID 9925057
- [Background] Tappero JW, Bradford WZ, Agerton TB, Hopewell P, Reingold AL, Lockman S, Oyewo A, Talbot EA, Kenyon TA, Moeti TL, Moffat HJ, Peloquin CA. Serum concentrations of antimycobacterial drugs in patients with pulmonary tuberculosis in Botswana. Clin Infect Dis. 2005 Aug 15;41(4):461-9. doi: 10.1086/431984. Epub 2005 Jul 8. PMID 16028152
- [Background] Grosset J, Leventis S. Adverse effects of rifampin. Rev Infect Dis. 1983 Jul-Aug;5 Suppl 3:S440-50. doi: 10.1093/clinids/5.supplement_3.s440. PMID 6356277
- [Background] Brindle R, Odhiambo J, Mitchison D. Serial counts of Mycobacterium tuberculosis in sputum as surrogate markers of the sterilising activity of rifampicin and pyrazinamide in treating pulmonary tuberculosis. BMC Pulm Med. 2001;1:2. doi: 10.1186/1471-2466-1-2. PMID 11737875
- [Background] Mitchison DA. Assessment of new sterilizing drugs for treating pulmonary tuberculosis by culture at 2 months. Am Rev Respir Dis. 1993 Apr;147(4):1062-3. doi: 10.1164/ajrccm/147.4.1062. No abstract available. PMID 8466107
- [Background] Mitchison DA. Modern methods for assessing the drugs used in the chemotherapy of mycobacterial disease. Soc Appl Bacteriol Symp Ser. 1996;25:72S-80S. No abstract available. PMID 8972122
- [Background] Jindani A, Aber VR, Edwards EA, Mitchison DA. The early bactericidal activity of drugs in patients with pulmonary tuberculosis. Am Rev Respir Dis. 1980 Jun;121(6):939-49. doi: 10.1164/arrd.1980.121.6.939. No abstract available. PMID 6774638
- [Background] Wallis RS, Perkins MD, Phillips M, Joloba M, Namale A, Johnson JL, Whalen CC, Teixeira L, Demchuk B, Dietze R, Mugerwa RD, Eisenach K, Ellner JJ. Predicting the outcome of therapy for pulmonary tuberculosis. Am J Respir Crit Care Med. 2000 Apr;161(4 Pt 1):1076-80. doi: 10.1164/ajrccm.161.4.9903087. PMID 10764293
- [Background] Burman WJ. The hunt for the elusive surrogate marker of sterilizing activity in tuberculosis treatment. Am J Respir Crit Care Med. 2003 May 15;167(10):1299-301. doi: 10.1164/rccm.2302003. No abstract available. PMID 12738594
- [Background] Jindani A, Dore CJ, Mitchison DA. Bactericidal and sterilizing activities of antituberculosis drugs during the first 14 days. Am J Respir Crit Care Med. 2003 May 15;167(10):1348-54. doi: 10.1164/rccm.200210-1125OC. Epub 2003 Jan 6. PMID 12519740
- [Background] Sirgel FA, Fourie PB, Donald PR, Padayatchi N, Rustomjee R, Levin J, Roscigno G, Norman J, McIlleron H, Mitchison DA. The early bactericidal activities of rifampin and rifapentine in pulmonary tuberculosis. Am J Respir Crit Care Med. 2005 Jul 1;172(1):128-35. doi: 10.1164/rccm.200411-1557OC. Epub 2005 Apr 1. PMID 15805182
- [Background] Hafner R, Cohn JA, Wright DJ, Dunlap NE, Egorin MJ, Enama ME, Muth K, Peloquin CA, Mor N, Heifets LB. Early bactericidal activity of isoniazid in pulmonary tuberculosis. Optimization of methodology. The DATRI 008 Study Group. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):918-23. doi: 10.1164/ajrccm.156.3.9612016. PMID 9310014
- [Background] Desjardin LE, Perkins MD, Wolski K, Haun S, Teixeira L, Chen Y, Johnson JL, Ellner JJ, Dietze R, Bates J, Cave MD, Eisenach KD. Measurement of sputum Mycobacterium tuberculosis messenger RNA as a surrogate for response to chemotherapy. Am J Respir Crit Care Med. 1999 Jul;160(1):203-10. doi: 10.1164/ajrccm.160.1.9811006. PMID 10390401
- [Background] Peloquin CA. Pharmacological issues in the treatment of tuberculosis. Ann N Y Acad Sci. 2001 Dec;953:157-64. doi: 10.1111/j.1749-6632.2001.tb11374.x. PMID 11795409
- [Background] Ribeiro-Rodrigues R, Resende Co T, Johnson JL, Ribeiro F, Palaci M, Sa RT, Maciel EL, Pereira Lima FE, Dettoni V, Toossi Z, Boom WH, Dietze R, Ellner JJ, Hirsch CS. Sputum cytokine levels in patients with pulmonary tuberculosis as early markers of mycobacterial clearance. Clin Diagn Lab Immunol. 2002 Jul;9(4):818-23. doi: 10.1128/cdli.9.4.818-823.2002. PMID 12093679
- [Background] Quaedvlieg V, Henket M, Sele J, Louis R. Cytokine production from sputum cells in eosinophilic versus non-eosinophilic asthmatics. Clin Exp Immunol. 2006 Jan;143(1):161-6. doi: 10.1111/j.1365-2249.2005.02968.x. PMID 16367947
- [Background] Colombo C, Costantini D, Rocchi A, Cariani L, Garlaschi ML, Tirelli S, Calori G, Copreni E, Conese M. Cytokine levels in sputum of cystic fibrosis patients before and after antibiotic therapy. Pediatr Pulmonol. 2005 Jul;40(1):15-21. doi: 10.1002/ppul.20237. PMID 15858808
- [Background] Husson MO, Wizla-Derambure N, Turck D, Gosset P, Wallaert B. Effect of intermittent inhaled tobramycin on sputum cytokine profiles in cystic fibrosis. J Antimicrob Chemother. 2005 Jul;56(1):247-9. doi: 10.1093/jac/dki179. Epub 2005 Jun 2. PMID 15932936
- [Background] Casarini M, Ameglio F, Alemanno L, Zangrilli P, Mattia P, Paone G, Bisetti A, Giosue S. Cytokine levels correlate with a radiologic score in active pulmonary tuberculosis. Am J Respir Crit Care Med. 1999 Jan;159(1):143-8. doi: 10.1164/ajrccm.159.1.9803066. PMID 9872832
- [Background] Verver S, Warren RM, Beyers N, Richardson M, van der Spuy GD, Borgdorff MW, Enarson DA, Behr MA, van Helden PD. Rate of reinfection tuberculosis after successful treatment is higher than rate of new tuberculosis. Am J Respir Crit Care Med. 2005 Jun 15;171(12):1430-5. doi: 10.1164/rccm.200409-1200OC. Epub 2005 Apr 14. PMID 15831840
- [Background] van Rie A, Victor TC, Richardson M, Johnson R, van der Spuy GD, Murray EJ, Beyers N, Gey van Pittius NC, van Helden PD, Warren RM. Reinfection and mixed infection cause changing Mycobacterium tuberculosis drug-resistance patterns. Am J Respir Crit Care Med. 2005 Sep 1;172(5):636-42. doi: 10.1164/rccm.200503-449OC. Epub 2005 Jun 9. PMID 15947286
- [Background] Kibiki GS, Mulder B, Dolmans WM, de Beer JL, Boeree M, Sam N, van Soolingen D, Sola C, van der Zanden AG. M. tuberculosis genotypic diversity and drug susceptibility pattern in HIV-infected and non-HIV-infected patients in northern Tanzania. BMC Microbiol. 2007 May 31;7:51. doi: 10.1186/1471-2180-7-51. PMID 17540031
- [Derived] Aarnoutse RE, Kibiki GS, Reither K, Semvua HH, Haraka F, Mtabho CM, Mpagama SG, van den Boogaard J, Sumari-de Boer IM, Magis-Escurra C, Wattenberg M, Logger JGM, Te Brake LHM, Hoelscher M, Gillespie SH, Colbers A, Phillips PPJ, Plemper van Balen G, Boeree MJ; PanACEA Consortium. Pharmacokinetics, Tolerability, and Bacteriological Response of Rifampin Administered at 600, 900, and 1,200 Milligrams Daily in Patients with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e01054-17. doi: 10.1128/AAC.01054-17. Print 2017 Nov. PMID 28827417